CLINICAL TRIAL: NCT05177731
Title: Comparing the Efficacy and Safety of Venetoclax Combined With Decitabine Versus Conventional "7+3" Induction Chemotherapy of Acute Myeloid Leukemia in Young Adults
Brief Title: Venetoclax + Decitabine vs. "7+3" Induction Chemotherapy in Young AML
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chen Suning (Other)
Responsible Party: Sponsor-Investigator, Chen Suning, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-AML02
Record Dates: First submitted 2021-12-27; First posted 2022-01-05 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: AML, Adult; Chemotherapy Effect
Keywords: Venetoclax, AML, young, induction therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Decitabine; Injections; Cytarabine; Idarubicin; gilteritinib

STUDY DESIGN:
Intervention Model Description: De novo adult AML patients randomly assigned to two induction treatment groups: venetoclax+decitabine group and conventional idarubicin(12mg/m2)+cytarabine group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational ( venetoclax, decitabine) (Experimental): Randomized participants will receive induction as decitabine on days 1-5 and venetoclax daily on days 1-28.
  Second Induction (if not reach complete remission, but the percentage of blaste cells in bone marrow decreased by more than 50%):Re-induction with pre-induction therapy.
  Consolidation: If patients with favorable risk and MRD (Minimal Residual Disease) negative or refuse to allo-HSCT (Hematopoietic stem-cell transplantation), intermediate-dose (2g/m2 q12h days 1-3) for 4 cycles. If patients with intermediate or poor risk or favorable risk but MRD positive, intermediate-dose cytarabine for 1-2 cycles and follow up with allo-HSCT.
  For patients with FLT3 mutation, gilteritinib can be combined with the follow-up treatment after the end of initial induction.
  Interventions: Drug: Venetoclax; Drug: Decitabine for Injection; Drug: Gilteritinib
- Standard of Care (Conventional Induction "7+3") (Experimental): Randomized participants will receive cytarabine and idarubicin per standard of care as follows:
  Induction: cytarabine on days 1-7 and idarubicin (12mg/m2) on days 1-3 .
  Second Induction (if not reach complete remission, but the percentage of blaste cells in bone marrow decreased by more than 50%): Re-induction with pre-induction therapy.
  Consolidation: If patients with favorable risk and MRD negative or refuse to allo-HSCT, intermediate-dose cytarabine (2g/m2 q12h days 1-3) for 4 cycles. If patients with intermediate or poor risk or favorable risk but MRD positive, intermediate-dose cytarabine for 1-2 cycles and follow up with allo-HSCT.
  For patients with FLT3 mutation, gilteritinib can be combined with the follow-up treatment after the end of initial induction.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Gilteritinib

INTERVENTIONS:
Drug: Venetoclax — Orally by mouth
  Other Names: Venclexta
  Arms: Investigational ( venetoclax, decitabine)
Drug: Decitabine for Injection — Intravenous infusion
  Arms: Investigational ( venetoclax, decitabine)
Drug: Cytarabine — Intravenous infusion
  Other Names: Ara-C
  Arms: Standard of Care (Conventional Induction "7+3")
Drug: Idarubicin — Intravenous infusion
  Other Names: IDA
  Arms: Standard of Care (Conventional Induction "7+3")
Drug: Gilteritinib — Orally by mouth
  Other Names: XOSPATA

SUMMARY:
This research is being done to assess the therapeutic efficacy and safety of a promising (venetoclax and decitabine) versus conventional "7+3"chemotherapy in induction young patients with acute myeloid leukemia.

This study involves the following:

Venetoclax and decitabine (investigational combination) Cytarabine and idarubicin (per standard of care)

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 2 randomized clinical trial to compare the therapeutic efficacy and safety of venetoclax and decitabine to the conventional induction chemotherapy (7+3 regimen) among fit, young adults with newly diagnosed acute myeloid leukemia (AML).

Conventional induction chemotherapy with idarubicin and cytarabine is the standard of induction chemotherapy for acute myeloid leukemia (AML).

The FDA has approved the combination therapy of venetoclax and decitabine for elderly (> 60 year old) patients with newly diagnosed AML not eligible for intensive chemotherapy. Venetoclax is an inhibitor of BCL-2 (B-cell lymphoma 2, a protein that initiates tumor growth, disease progression, and drug resistance), which can lead to cancer cell death. Decitabine, a demethylation agent, has the potential to synergically target leukemia stem cell populations when combined with venetoclax as its homologous drug azacytidine.

Participants will be randomly assigned to one of the different induction groups and followed with either consolidation chemotherapy or allogeneic hematopoietic stem cell transplantation after remission. After completion of study treatment, participants are followed up every 3 to 6 months for up to 2 years.

It is expected that about 188 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 59 > =Age (years) >= 18;
2. Newly diagnosed as AML patients according to World Health Organization (WHO) 2016 classification;
3. Patients have not received prior therapy for AML (except hydroxyurea and Ara-C<1.0g/d);
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0,1, 2 ;
5. Liver function: Total bilirubin ≦3 upper limit of normal (ULN); aspartate aminotransferase (AST) ≦3 ULN; alanine aminotransferase (ALT)≦3 ULN(except extramedullary infiltration of leukemia)
6. Renal function：Ccr（Creatinine Clearance Rate） ≧30 ml/min;
7. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Acute promyeloid leukemia；
2. AML with central nervous system (CNS) infiltration；
3. Patients have received prior hypomethylating agents (HMA) therapy for myelodysplastic syndrome (MDS) and progressed to AML；
4. HIV infection;
5. Patients with severe heart failure (grade 3-4) ;
6. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to: a) Uncontrolled and/or active systemic infection (viral, bacterial or fungal); b) Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. c) An active second cancer that requires treatment within 6 months of study entry
7. Patients deemed unsuitable for enrolment by the investigator;
8. Patients willing to receive intensive induction chemotherapy
9. Female who are pregnant, breast feeding or childbearing potential without a negative urine pregnancy test at screen；
10. Patients reject to participate in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From randomization to 2 cycles of induction before consolidation therapy（100 days）
  Complete remission/complete remission with incomplete count recovery/Morphologic Leukemia Free State

SECONDARY OUTCOMES:
Incidence of severe infection (>=grade 3 ) | From randomization to 2 cycles of induction before consolidation therapy（100 days）
  Assessed using CTCAE 5
Duration of myelosuppression | From randomization to 2 cycles of induction before consolidation therapy（100 days）
  The duration of absolute value of peripheral blood neutrophils <0.5×10^9/L and platelet count <50×10^9/L during myelosuppression.
Event free survival | From the time from randomization to time for up to 2 years
  Events include progressive disease, relapse, changes in treatment regimens, fatal or intolerable side effects and any death.
Overall survival | From the time from randomization to time for up to 2 years
  Overall survival
Rate of Minimal Residual Disease (MRD) negativity | From randomization to 2 cycles of induction before consolidation therapy（100 days）
  Percentage of participants who converted to MRD < 10^-3 before initiation of consolidation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Lu J, Xue SL, Wang Y, He XF, Hu XH, Miao M, Zhang Y, Tang ZX, Xie JD, Yang XF, Xu MZ, Shen YY, Du F, Wu Q, Xue MX, Wang Y, Deng AL, Dou XQ, Xu Y, Dai HP, Wu DP, Chen SN. Venetoclax and decitabine vs intensive chemotherapy as induction for young patients with newly diagnosed AML. Blood. 2025 May 29;145(22):2645-2655. doi: 10.1182/blood.2024027217. PMID 40009498
- [Derived] Waclawiczek A, Leppa AM, Renders S, Stumpf K, Reyneri C, Betz B, Janssen M, Shahswar R, Donato E, Karpova D, Thiel V, Unglaub JM, Grabowski S, Gryzik S, Vierbaum L, Schlenk RF, Rollig C, Hundemer M, Pabst C, Heuser M, Raffel S, Muller-Tidow C, Sauer T, Trumpp A. Combinatorial BCL2 Family Expression in Acute Myeloid Leukemia Stem Cells Predicts Clinical Response to Azacitidine/Venetoclax. Cancer Discov. 2023 Jun 2;13(6):1408-1427. doi: 10.1158/2159-8290.CD-22-0939. PMID 36892565